CLINICAL TRIAL: NCT03813433
Title: Discoloration After Revascularization Using Calcium Phosphosilicate Based Bioceramic vs Mineral Trioxide Aggregate in Necrotic Immature Permanent Anterior Teeth: A Randomized Clinical Trial
Brief Title: Discoloration of Endosequence and Mineral Trioxde Aggregate in Revascularization of Necrotic Immature Permanent Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Tarek Bartaw, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pedodontic department cairo
Record Dates: First submitted 2019-01-14; First posted 2019-01-23 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-09

CONDITIONS: Pulp Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enosequence (Experimental): 3-4 mm of Endosequence will be applied over the blood clot in group I. Material will be packed using condenser with light pressure. Periapical radiograph will be taken to ensure coronal seal in the second visit of revascularization
  Interventions: Other: Revascularization
- Mineral Trioxide Aggregate (Active Comparator): 3-4 mm of Mineral Trioxide Aggregate will be applied over the blood clot in group I. Material will be packed using condenser with light pressure. Periapical radiograph will be taken to ensure coronal seal in the second visit of revascularization
  Interventions: Other: Revascularization

INTERVENTIONS:
Other: Revascularization — a procedure used to regenerate pulp dentin complex that restores the functional properties of this immature anterior teeth, prevent and resolves apical periodontitis
  Other Names: pulp regeneration

SUMMARY:
the objective of this study is to evaluate post operative pain after using Endosequence versus Mineral Trioxide Aggregate as coronal plug material in revascularization of non vital immature anterior teeth

DETAILED DESCRIPTION:
The treatment of immature young permanent anterior teeth is challenging because in addition of the need of elimination of bacterial infection; the lack of natural apical constriction against which a suitable filling material can be placed is considered the main problem.

In the past many different treatments have been proposed for immature permanent teeth with necrotic pulps such as:Custom fitting of filling materials like gutta percha, Periapical surgeries, apexification. The disadvantages of these treatments are: the compromised Crown/root ratio, possibility of vertical fracture.

Pulp revascularization is dependent on the ability of residual pulp and apical and periodontal stem cells to differentiate. These cells have the ability to generate a highly vascularized and rich living tissue.

MTA was chosen as coronal seal to be placed over the blood clot due its a biocompatibility, bio-inductivity. However, the disadvantages of MTA are: discoloration of the coronal dentine when placed in the canal and the difficult handling properties.

Recently, a new bioceramic material has been introduced to the market, namely, EndoSequence which is bioactive, has antibacterial activity, less cytotoxic effect and similar antimicrobial properties, maintain color stability of the tooth when compared to MTA

ELIGIBILITY:
Inclusion Criteria:

* Age of patient range from 8-14 y.
* Patients are free from any systemic diseases that may hinder the normal healing process.
* Non vital permanent anterior teeth with open apex.
* Pulp space not needed for post and core for final restoration.
* Compliant patient/parent.

Exclusion Criteria:

* Patients having allergy to medicaments and antibiotics necessary to complete the procedure.
* Tooth with vital pulp or complete root formation.
* Teeth with internal or external root resorption.
* Un-cooperative patients

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
discoloration | 1 month
  Asking patient question (Binary:present or absent)
discoloration | 3 months
  Asking patient question (Binary:present or absent)
dicoloration | 6 months
  Asking patient question (Binary:present or absent)
discoloration | 9 months
  Asking patient question (Binary:present or absent)
discoloration | 12months
  Asking patient question (Binary:present or absent)

SECONDARY OUTCOMES:
post operative pain | 1,3, 6, 9 and 12 months
  asking the patient (Binary: present or Absent)
color stability | 1,3, 6, 9 and 12 months
  Operator and supervisor evaluation (Using shade guide)
Pain on percussion | 1,3, 6, 9 and 12 months
  Assessed by back of the mirror (Binary: present or absent)
Swelling | 1,3, 6, 9 and 12 months
  assessed by visual examination (Binary:present or absent)
Sinus or fistula | 1,3, 6, 9 and 12 months
  assessed by visual examination (Binary:present or absent)
Root lengthening | 6 and 12 months
  assessed radiographically (DIGORA® for Windows software)